CLINICAL TRIAL: NCT03643497
Title: Population Pharmacokinetics of Meropenem and Linezolid in Children With Severe Infectious Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shandong University (Other); Hopital Universitaire Robert-Debre (Other); Rennes University Hospital (Other)
Responsible Party: Principal Investigator, Adong Shen, Deputy Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCH_PPK004
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Children；Infection
MeSH Terms: interventions — Anti-Infective Agents; Meropenem; Linezolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Biospecimen Retention: Samples With DNA — whole blood and plasma and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with the usage of anti-infective drugs: Children received meropenem or linezolid monotherapy in the treatment of seven infectious diseases
  Interventions: Drug: anti-infective drugs

INTERVENTIONS:
Drug: anti-infective drugs — According to the models of population pharmacokinetics, the investigators and want to correlate use of antibiotics with treatment effectiveness and safety in children
  Other Names: meropenem; linezolid

SUMMARY:
This study is based on the hypothesis that the pharmacokinetics of meropenem and linezolid in severe infectious children are different from mild infectious children and adults. The investigators aim to study the population pharmacokinetics of children receiving the meropenem and linezolid for treatment of severe infectious diseases. In this study, the investigators will detect drug concentration in plasma and cerebrospinal fluid by using residual blood samples of blood and cerebrospinal fluid gas analysis and other clinical tests and employ computers for constructing population pharmacokinetic models. In addition, the investigators also want to correlate use of meropenem and linezolid with treatment effectiveness and incidence of adverse effects in children. This novel knowledge will allow better and more rational approaches to the treatment of severe infectious diseases in children. It will also set the foundation for further studies to improve anti- infective drug therapies for severe infectious children.

DETAILED DESCRIPTION:
1.Establish population pharmacokinetic (PPK) models of meropenem and linezolid in severe infectious children by nonlinear mixed effect modeling (NONMEM).

1. At different time point after meropenem or linezolid administration, plasma and/or cerebrospinal fluid samples of 100 children will be collected from pediatric intensive care unit (PICU) for each drug. The clinical information includes demography, medication, concentration data, blood biochemical parameters and so on.
2. Plasma and cerebrospinal fluid samples will be tested by high performance liquid chromatography (HPLC).
3. PPK models of meropenem and linezolid will be established by NONMEM program.
4. The reliability and stability of the PPK model will be evaluated by 1000 times of Bootstrap procedure and normalized predictive distribution error(NPDE).

2. Evaluation of the clinical feasibility and safety of individualized dosing.

1. According the results of PPK models, the investigators will use dosages recommended in models to cure severe infectious children in prospective studies. For antibiotic drug, 50 children will be collected.
2. The investigators will compare the therapeutic effects and safety between children with conventional therapies and children with individualized therapies in severe infectious diseases, including proportions of children with effective drug concentration, improvement speed of children, liver and kidney functions of children, adverse reactions of drugs and so on

ELIGIBILITY:
Inclusion Criteria:

* Children (0-18 years old) with anti-infective therapy against severe infectious diseases.
* The anti-infective therapy includes meropenem and linezolid commonly used in children with infectious diseases,
* Children severe infectious diseases include severe pneumonia, sepsis, purulent meningitis and other diseases with severe infection.
* Informed consent signed by the parents and/or guardians

Exclusion Criteria:

* Anti-infective drugs aren't involved in the therapies of children.
* It is unable to provide complete medical records or the current condition cannot accept the study process.
* Patients are allergic to meropenem or linezolid.
* Parents and/or guardians do not agree to participate in this study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Severe infectious children with anti-infectious therapies
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | up to 4 weeks
  Cmax is a term used in pharmacokinetics refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose

SECONDARY OUTCOMES:
time to achieve maximum concentration (Tmax) | up to 4 weeks
  Tmax is the term used in pharmacokinetics to describe the time at which the Cmax is observed
absorption rate constant (ka) | up to 4 weeks
  Ka is the rate constant of drug absorption
elimination rate constant (kel) | up to 4 weeks
  The elimination rate constant is a value used in pharmacokinetics to describe the rate at which a drug is removed from the system
half-life (t1/2) | up to 4 weeks
  Half-life is the time required for a quantity to reduce to half its initial value

CONTACTS AND LOCATIONS:
Overall Officials: Shen A-Dong, Master, Principal Investigator — Beijing Children's Hospital of Capital Medical University; Qi Yu-Jie, Master, Study Director — Beijing Children's Hospital of Capital Medical University; Zhao Wei, Doctor, Study Director — Children's Hospital of Hebei Province;Shandong Provincial Qianfoshan Hospital
Locations (1):
- Beijing Children's Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Jacqz-Aigrain E, Leroux S, Zhao W, van den Anker JN, Sharland M. How to use vancomycin optimally in neonates: remaining questions. Expert Rev Clin Pharmacol. 2015;8(5):635-48. doi: 10.1586/17512433.2015.1060124. Epub 2015 Aug 4. PMID 26289222
- [Result] Ramos-Martin V, Johnson A, Livermore J, McEntee L, Goodwin J, Whalley S, Docobo-Perez F, Felton TW, Zhao W, Jacqz-Aigrain E, Sharland M, Turner MA, Hope WW. Pharmacodynamics of vancomycin for CoNS infection: experimental basis for optimal use of vancomycin in neonates. J Antimicrob Chemother. 2016 Apr;71(4):992-1002. doi: 10.1093/jac/dkv451. Epub 2016 Jan 10. PMID 26755499
- [Result] Zhao W, Hill H, Le Guellec C, Neal T, Mahoney S, Paulus S, Castellan C, Kassai B, van den Anker JN, Kearns GL, Turner MA, Jacqz-Aigrain E; TINN Consortium. Population pharmacokinetics of ciprofloxacin in neonates and young infants less than three months of age. Antimicrob Agents Chemother. 2014 Nov;58(11):6572-80. doi: 10.1128/AAC.03568-14. Epub 2014 Aug 25. PMID 25155587
- [Derived] Wang Z, Bi J, You D, Tang Y, Liu G, Yu J, Jin Z, Jiang T, Tian X, Qi H, Dong L, Dong L, Zhang Q, Zhao W, Shen A. Improving the efficacy for meropenem therapy requires a high probability of target attainment in critically ill infants and children. Front Pharmacol. 2022 Oct 5;13:961863. doi: 10.3389/fphar.2022.961863. eCollection 2022. PMID 36278190
- [Derived] Wang ZM, Chen XY, Bi J, Wang MY, Xu BP, Tang BH, Li C, Zhao W, Shen AD. Reappraisal of the Optimal Dose of Meropenem in Critically Ill Infants and Children: a Developmental Pharmacokinetic-Pharmacodynamic Analysis. Antimicrob Agents Chemother. 2020 Jul 22;64(8):e00760-20. doi: 10.1128/AAC.00760-20. Print 2020 Jul 22. PMID 32513801